CLINICAL TRIAL: NCT03032848
Title: Randomized, Blinded Trial Comparing Vaginal Estrogens on Pelvic Organ Prolapse Patients
Brief Title: Vaginal Estrogens Comparative Trial on Pelvic Organ Prolapse Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Elisa Chicareli Pinhat, Doctor, Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 23286013.7.0000.0096; 475.622 (Registry Identifier: Opinion Number)
Record Dates: First submitted 2017-01-20; First posted 2017-01-26 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Vaginitis Atropic; Pelvic Organ Prolapse; Endometrial Hyperplasia
MeSH Terms: conditions — Atrophic Vaginitis; Pelvic Organ Prolapse; Endometrial Hyperplasia | interventions — Estrogens, Conjugated (USP); promestriene; Estriol

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conjugated Estrogen Group (Active Comparator): use of 1 gram per day
  Interventions: Drug: Promestriene; Drug: Estriol; Drug: Vaginal Moisturizer - Cream
- Promestriene Group (Active Comparator): use of 1 gram per day
  Interventions: Drug: Conjugated Estrogen; Drug: Estriol; Drug: Vaginal Moisturizer - Cream
- Estriol Group (Active Comparator): use of 1 gram per day
  Interventions: Drug: Conjugated Estrogen; Drug: Promestriene; Drug: Vaginal Moisturizer - Cream
- Vaginal Moisturizer Cream (Placebo Comparator): use of 1 gram per day
  Interventions: Drug: Conjugated Estrogen; Drug: Promestriene; Drug: Estriol

INTERVENTIONS:
Drug: Conjugated Estrogen — use of 1 gram per day
  Other Names: Premarin
  Arms: Estriol Group; Promestriene Group; Vaginal Moisturizer Cream
Drug: Promestriene — use of 1 gram per day
  Other Names: Colpotrofine
  Arms: Conjugated Estrogen Group; Estriol Group; Vaginal Moisturizer Cream
Drug: Estriol — use of 1 gram per day
  Other Names: Stelle
  Arms: Conjugated Estrogen Group; Promestriene Group; Vaginal Moisturizer Cream
Drug: Vaginal Moisturizer - Cream — use of 1 gram per day
  Other Names: Vagidrat
  Arms: Conjugated Estrogen Group; Estriol Group; Promestriene Group

SUMMARY:
To evaluate the difference of three vaginal estrogens creams comparative with placebo on improvement of hormonal cytology, local and systemic climacteric complaints, as well as its endometrial security.

ELIGIBILITY:
Inclusion Criteria:

* post menopause women
* normal oncotic cytology and mammogram
* any grade of pelvic organ prolapse with surgery indication and ultrasound with endometrium measure less than 5 mm

Exclusion Criteria:

* vaginal bleeding
* hormonal replacement on the past three months
* renal or hepatic desease
* porfiria
* past venous thromboembolism; ulcerated prolapse

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-26 (Actual)

PRIMARY OUTCOMES:
Evaluate the histopathological effects on endometrium after each treatment | 48 days
  Compare the histopathological results after treatment on each group and among each other
Compare the endometrial thickness measured by ultrassound after each treatment | 48 days
  Compare the endometrial ultrasound measurement before and after treatment in each group, and among each other

SECONDARY OUTCOMES:
Evaluate the changes of maturation index (Meisels Index) after each treatement | 48 days
  Compare the changes on Meisels Index after each treatment and among each other
Evaluate the changes on climacteric complaints after each treatment | 48 days
  Compare the changes on systemic and genital complaints after each treatment, and among each other

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Management of symptomatic vulvovaginal atrophy: 2013 position statement of The North American Menopause Society. Menopause. 2013 Sep;20(9):888-902; quiz 903-4. doi: 10.1097/GME.0b013e3182a122c2. PMID 23985562
- [Derived] Taithongchai A, Johnson EE, Ismail SI, Barron-Millar E, Kernohan A, Thakar R. Oestrogen therapy for treating pelvic organ prolapse in postmenopausal women. Cochrane Database Syst Rev. 2023 Jul 11;7(7):CD014592. doi: 10.1002/14651858.CD014592.pub2. PMID 37431855